CLINICAL TRIAL: NCT04656327
Title: Oral Health Status in Care-dependent Community Dwelling Elders: a Cross-sectional Study in Zurich
Brief Title: Oral Health Status in Care-dependent Community Dwelling Elders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Murali Srinivasan, Professor, University of Zurich
Other Study IDs: UZH_ABS_2020_2
Record Dates: First submitted 2020-11-17; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Oral-health; Nutritional Status

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non interventional group: Community-dwelling elders dependent for care
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this study. It is a cross-section study evaluating the oral health and nutritional statuses of community-dwelling elders dependent for care for their activities of daily living.

SUMMARY:
The primary aim of this cross-sectional survey in Zurich is to assess the oral health status (OHS), Oral Health Related Quality of Life (OHRQoL), and the nutritional status (NS) of community-dwelling elders dependent for care. The secondary objective of this study evaluates whether the OHS, OHRQoL and NS are influenced by cognitive status, level of dependency, socio-economic status and level of education. The tertiary objective is to assess whether the quality of nutritional uptake (refrigerator content) by the community-dwelling elders dependent for care is influenced by OHS/function, level of dependency, cognitive impairment, socio-economic status or level of education and the proximity and/or access to food sources (supermarkets).

DETAILED DESCRIPTION:
Aim: The aim of this cross-sectional study is to assess the oral health status, Oral Health Related Quality of Life, and the nutritional status of community-dwelling elderly adults requiring care for their activities of daily living.

Methods:

Community dwelling elders residing in their homes but receiving out-patient care will be recruited in this study. Participants will receive a detailed oral examination at their residences. Their oral health status and oral function will be evaluated according to the following indices: DMF(T), plaque index (Plx), gingival index (GIx), community periodontal index for treatment needs (CPITN), xerostomia inventory (XI), brushing habits, denture calculus index (DCI), Denture Assessment (Marxkors Criteria), chewing efficiency (CE) and maximum bite force (MBF). The quality of oral care will be assessed by the use and condition of the prevalent oral hygiene tools according to the Toothbrush wear rate (TBWR). Furthermore, the Quality of Life (QoL) and Oral Health Related Quality of Life (OHRQoL) will be measured with the Oral health impact profile 14 items (OHIP-14) and EuroQol-5D (EQ-5D). Finally, the nutritional status of these care-dependent elders will be recorded with the mini nutritional assessment (MNA) as well as the recording their refrigerator content along with a 24-hour diet chart.

Discussion:

The population is ageing worldwide and teeth are being retained to an advanced age. Oral health however declines, in elders dependent for care, due to age associated complications including, multi morbidity, poly-pharmacy, cognitive and physical impairments. As a consequence, edentulous state prevails at a later age. Prevention and oral hygiene maintenance become difficult in these elders and even more complex in those who are rehabilitated with prosthetic reconstructions. Oral hygiene and care is very important in these individuals to prevent and intervene the disease process. Tooth loss combined with cognitive decline, frailty and other age-associated complications may lead to malnutrition. This study hopes to provide a reliable evaluation of the current oral health and nutritional status of elderly people living in the community and are dependent for care in an industrialised country. These data are considered cardinal and imperative for both government policies in terms of preventive programs, health educations, as well as for the organisation providing these care services.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Living in their residence in the canton of Zurich but dependent for care for their Activities of Daily Living (ADLs)

Exclusion Criteria:

1. Not willing or able to sign informed consent or not given by the caregiver/guardian.
2. Age < 65 years
3. Non-responsive / not cooperative for examination

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly population living in the canton of Zurich, who are care-dependent and community- dwelling receiving out-patient care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-26 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | Day 1
  Sillness and Löe Plaque index: The index measures the state of oral hygiene based on the amount of soft and mineralised debris present on the 6 indexed teeth (teeth no. 16, 12, 24, 36, 32 & 44). The following grades will be allotted to the teeth based on the observed debris state on its four surfaces (Labial/Buccal, Mesial, Distal & Palatal/Lingual):
  0- No plaque
  1. A film of plaque adhering to the free gingival margin (plaque detectable only by probing)
  2. Moderate accumulation of plaque (plaque perceivable by naked eye and interdental space is free).
  3. Abundance of plaque (Interdental space is filled with plaque) x- Tooth not present. The four scores per tooth are summed and an average per tooth is calculated for that tooth. Then the mean of all the individual average scores of the examined teeth is calculated. This number gives us the plaque index for the patient.
Gingival index | Day 1
  Löe and Silness Gingival Index : The index measures the degree of inflammation of the gingiva on the 6 indexed teeth (teeth no. 16, 12, 24, 36, 32 & 44). The following grades will be allotted to the teeth based on the bleeding present after a careful probing of the gingival sulcus:
  0- Normal gingiva (No inflammation, no discolouration, no bleeding, no loss of stippling)
  1. Low inflammation (slight color change, no bleeding)
  2. Moderate inflammation (redness, oedema, bleeding on probing, loss of stippling).
  3. Severe inflammation (redness, oedema, tendency to spontaneously bleed, ulceration, loss of stippling) x- Tooth not present The four scores per tooth are summed and an average per tooth is calculated for that tooth. Then the mean of all the individual average scores of the examined teeth is calculated. This number gives us the gingival index for the patient.
DMF(T) | Day 1
  Decayed, Missing, Filled (Teeth) index: Each tooth present in the mouth will be graded as either decayed, missing or filled. Then all the numbers are added up to give us the DMF(T) status of the patient.
CPITN index | Day 1
  This index measures the state of the oral health in terms of periodontal disease and the treatment needs for the patient.
  All the teeth are examined and the most affected tooth per sextant is awarded a score. The following scores are possible for the teeth examined:
  0- healthy (No bleeding on probing, no marginal irritation, no pockets): No treatment.
  1. No pockets, Bleeding on Probing, no calculus, no overhangs. Treatment: Oral hygiene instructions (OHI)
  2. Pockets <3mm, sub gingival calculus present, and/or iatrogenic marginal irritations (overhanging restoration margins). Treatment: OHI, scaling and correction of overhangs.
  3. Deepest pockets between 4 and 5 mm. Treatment: OHI, Scaling and root planing.
  4. Probing depth >6 mm. Treatment: Scaling & root planing, and/or flap as required.
     * - furcation is involved and/or a total loss of attachment >7mm is present. Treatment: Full periodontal examinations of all sextants regardless of CPITN score.
Dentition Status | Day 1
  Assessment of status of dentition in the mouth. The examination will classify the edentulism present in the jaw as either completely edentate or partially dentate. And if Partially edentate, then the Kennedy's Classification will be applied to classify the partial edentulism present in the jaw.
  We will also examine if the edentulism present is rehabilitated with what type of prosthesis ( fixed dental prosthesis/removabnle dental prosthesis/Implant supported fixed dental prosthesis or implant supported removable dental prosthesis)
Denture Calculus index (DCI) | Day 1
  Denture calculus index measures the amount of soft and hard debris present on the removable dental prosthesis.
  The following grades are allotted based on the presence of the debris on the prosthesis:
  0- No visible plaque
  1. Plaque visible only by scrapping
  2. Moderate visible plaque
  3. Abundant plaque present
Maximum bite force (MBF) | Day 1
  Maximum bite force is measured using a bite force meter. The patient will be requested to bite on the bite force meter first on the right side. The patient will then be requested to do the same on the left side. Three observations will be recorded for each side. The mean of the maximum bite force from both sides will be calculated and used for the analysis.
Chewing function (CE) | Day 1
  Chewing function is measured using a bi-color chewing gum. The patient will chew on the chewing gums for 20 chewing cycles. The gum is flattened to a wafer thickness of 1 mm. Both sides of this wafer are scanned with a flat-bed photo scanner. The two images are brought together on a single frame using a photo software. This single image is then imported into a software (ViewGum). The software calculates the variance of hue (VoH) for each chewing gum. VoH is a numerical value and the lower the value better is the chewing efficiency.
  A visual subjective assessment (SA) of the chewing gums will also be performed. The following grades will be allotted:
  SA1- Chewing not mixed, only impressions of cusps are p[resent or the chewing appears folded without being mixed.
  SA2- Large parts of the chewing gums are mixed. SA3- Bolus slightly mixed but bits of unmixed original color still present. SA4- Bolus well mixed, but color not uniform. SA5- Bolus perfectly mixed with uniform color.
Oral health impact profile 14-items (OHIP-14) | Day 1
  OHIP-14 measures the Quality of life related to oral health. It is a subjective assessment which captures 7 dimensions (Functional limitation, Physical pain, Psychological discomfort, Physical disability, Psychological disability, Social disability and Handicap) by the means of 14- items. The participant must respond with a Likert scale-type response (4-Very often, 3-Often, 2-from time to time, 1- rarely, 0-Never). The lower the score, the better the Oral health related Quality of life (OHRQoL).
European Quality of Life - 5 Dimensions (EQ-5D) | Day 1
  EQ-5D measures the general health status not specific to a disease. There are 5 dimensions (Mobility, self care, usual activities, pain/discomfort, and anxiety/depressions). There is one question per dimension and a possible Likert scale response type with three options (1- No problems, 2-Some problems, 3-Too much problems). A score between 1 and 3 is given to each of the dimensions.
Xerostomia Inventory with 11-items (XI-11) | Day 1
  XI-11 assesses the xerostomia state of the participant. There are 11 questions in the inventory and the patient has the possibility to respond with a Likert-scale type response type (4-Very often, 3-Often, 2-from time to time, 1- rarely, 0-Never). The lower the score the better the index and shows the absence/reduced xerostomia.
Mini-Nutritional Assessment (MNA) | Day 1
  The MNA instrument measures the nutritional state of the patient and its primary targets are under- and malnutrition states. The instrument has a two-stage structure and anamnesis with 6 items with a further 12 items including two anthropometric measurements (upper arm circumference and calf circumference). The maximum score is 30 points. The scale is:
  17-23.5: risk for malnutrition <17: poor nutritional state
Refrigerator Content | Day 1
  In this, we will make a record of all the items present in the participants refrigerator. All the items present will be assessed for validity of expiry and nutritional values will be calculated based on the information present on the box/label.
Oral hygiene tools and maintenance | Day 1
  In this outcome, information on the frequency of the oral hygiene performed, the tools employed, condition of the oral hygiene tools present will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Murali Srinivasan, BDS, MDS, MBA, MAS, Principal Investigator — University of Zurich
Locations (1):
- Clinic of General, Special care, and Geriatric Dentistry, Center of Dental Medicine, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No